CLINICAL TRIAL: NCT05147766
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Heart Disease
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for Heart Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient efficacy seen in treated patients
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-017
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Congestive Heart Failure; Angina
Keywords: Angina; Congestive Heart Failure; stem cell treatment
MeSH Terms: conditions — Heart Failure; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of congestive heart failure and angina

DETAILED DESCRIPTION:
This patient funded trial aims to study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of congestive heart failure and angina. Patients will receive a single intravenous infusion of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease an autologous Effector cells (activated lymphocytes) treatment will be utilized created from the patient's own cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Congestive Heart Failure or Angina
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No